CLINICAL TRIAL: NCT06284837
Title: Secondary Access - FEmoral or Radial in Transcatheter Aortic Valve Implantation?
Acronym: SAFER-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Epworth Healthcare (Other); Cabrini Health (Other)
Responsible Party: Principal Investigator, Kawa Haji, Principal investigator, The Alfred
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HREC/99382/Alfred-2023
Record Dates: First submitted 2023-12-08; First posted 2024-02-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Valve Stenoses, Aortic
Keywords: TAVI; TAVR; transcatheter aortic valve replacement; transcatheter aortic valve implantation; aortic stenosis; vascular access; primary access; secondary access
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: SAFER-TAVI trial is a multicentre registry-nested, randomised controlled trial comparing transradial versus transfemoral secondary access in patients undergoing transfemoral TAVI for aortic valve disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radial secondary access (Active Comparator)
  Interventions: Other: Access site
- Femoral secondary access (Active Comparator)
  Interventions: Other: Access site

INTERVENTIONS:
Other: Access site — The SAFER-TAVI trial is randomized study comparing secondary access via a transradial versus transfemoral approach among patients undergoing transfemoral TAVI for aortic valve disease. Secondary access is gained along with primary access at the commencement of the TAVI procedure and is used for aortography before and after valve deployment and for assessment of the primary femoral access site after closure to confirm haemostasis. For patients assigned to radial access, the radial sheath will be removed using a radial band at the end of the procedure. For patients assigned to femoral access, the puncture site will be obtained under ultrasound guidance and fluoroscopic landmark identification. Unless contraindicated, the use of vascular closure devices will be recommended for all femoral cases. The choice of closure device is at the discretion of the operator. Catheters used in the access groups will be 5 or 6 French size at the discretion of the operator.

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a well-known safe and effective treatment for anatomically suitable patients with severe aortic stenosis (AS). Despite rapid improvements in TAVI technique and technology, vascular and bleeding complications from both primary and secondary access sites remain significant, with approximately 25% of access related complications thought to be related to secondary access. The transfemoral route remains the most common approach for primary access during TAVI due to proven safety and efficacy. Secondary access during TAVI, which is needed for angiographic guidance, has drawn little attention in randomised trials of TAVI. In coronary intervention, the radial approach is now preferred due to high quality evidence suggesting lower bleeding and vascular complications compared to the femoral approach. Whilst randomised control trials comparing radial vs femoral as secondary access are lacking in the TAVI setting, observational studies comparing the two secondary access routes have shown a lower risk of bleeding and vascular complications with radial compared to femoral access. A systematic review of all the major observational trials also suggests that radial access might reduce risk of bleeding, vascular complications, and even 30-day mortality, but these data are limited to observational trials and there are no randomised controlled data to confirm these findings. Accordingly, we aim to undertake a multicentre, randomised controlled trial among patients undergoing transfemoral TAVI to assess if radial secondary access is superior to femoral secondary access.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Undergoing transfemoral TAVI with any commercially available transcatheter heart valve
* Suitable radial and secondary femoral access

Exclusion Criteria:

* Primary arterial access via surgical cut-down
* Inadequate contralateral femoral artery access and/or bilateral radial artery access as determined by the interventional cardiologist
* Previously failed attempt to access bilateral radial arteries.
* Patient on hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
All clinically relevant bleeding and all vascular complications | 30 days
  The composite of all clinically relevant bleeding (defined as Bleeding Academic Research Consortium [BARC] type ≥2) and vascular complications (Valve Academic Research Consortium [VARC3] criteria) at 30 days.

SECONDARY OUTCOMES:
All clinically relevant bleeding (BARC ≥2), overall and by access site | 30 days
  Using BARC criteria
All vascular complications, overall and by access site | 30 days
  Using VARC-3 criteria
All-cause death | 30 days
  Using VARC-3 criteria
Stroke | 30 days
  Using VARC-3 criteria
Myocardial infarction | 30 days
  Using VARC-3 criteria
Major adverse cardiovascular events | 30 days
  The composite of cardiovascular death, non-fatal myocardial infarction and non-fatal stroke
Length of stay post-procedure | 30 days
  Length of stay post-procedure measured in time (days) from procedure to discharge
Overall procedure duration | 1 day
  TAVI procedure duration measured in time (minutes)
Radiation dose | 1 day
  Radiation dose measured as air kerma in milligrays
Conversion rate to alternative vascular access site | 30 days
  Conversion rate to alternative vascular access site
Tertiary site utilised to treat vascular complication | 30 days
  Tertiary site utilised to treat vascular complication
Failure to perform angiogram of primary access site at completion of TAVI | 1 day
  Failure to perform angiogram of primary access site at completion of TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Antony Walton, MBBS, Principal Investigator — The Alfred and Epworth Healthcare; Dion Stub, MBBS, PhD, Principal Investigator — The Alfred and Cabrini Health
Locations (3):
- Australia (3):
  - Alfred Health, Melbourne, Victoria
  - Epworth Healthcare, Melbourne, Victoria
  - Cabrini Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
Yes if ethics is approved